CLINICAL TRIAL: NCT06739031
Title: A Multi-center, Single-group Clinical Trial to Evaluate the Efficacy and Safety of Pulsed Electric Field (PEF) Ablation Devices in the Treatment of Lung Tumors
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Pulsed Electric Field Ablation Devices in the Treatment of Lung Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Energenx Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC-101
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEF Treatment (Experimental)
  Interventions: Device: PEF Treatment

INTERVENTIONS:
Device: PEF Treatment — PEF Energy ablation of lung tumors

SUMMARY:
The goal of this clinical trial is to verify the efficacy and safety of pulsed electric field (PEF) treatment of early-stage unreseectable non-small cell lung cancer(NSCLC) patients.

The main questions it aims to answer are:

* Safety of PEF treatment of early-stage unreseectable NSCLC patients.
* Locoregional control of ablated lesions.
* Survival and quality of life assessment of early-stage unreseectable NSCLC patients.

ELIGIBILITY:
Inclusion criteria (all requirements must be met at the same time):

1. Age ≥ 18 years old; 2. Pathological diagnosis of non-small cell lung cancer, with the maximum diameter of the tumor ≤ 3 cm and the number ≤ 3; 3. ECOG score ≤ 2 points; 5. According to the evaluation of the researcher, it is technically feasible to perform ablation treatment on the lesion; 6. The subject agrees to receive ablation treatment and signs the informed consent form.

Exclusion criteria (if any of the above conditions are met, the patient will be excluded):

1. The subject cannot tolerate or refuses general anesthesia;
2. Has a history of severe allergic reactions;
3. Has contraindications to bronchoscopy or refuses bronchoscopy;

5. Has active implants in the chest cavity or metal implants in the lung to be treated; 6. Uncorrectable coagulation abnormalities (INR>1.5 or APTT>1.5 ULN), with bleeding tendency; anticoagulant therapy and/or antiplatelet drugs are discontinued before ablation for no longer than the prescribed safety period; platelets <50×10^9/L; 7. Severe liver and kidney dysfunction, assessed by the researchers as unsuitable for inclusion; 8. Accompanied by infectious diseases that cannot be effectively controlled; 9. Subjects with other severe lung diseases (including severe interstitial pneumonia, pulmonary fibrosis, pulmonary fibrosis combined with emphysema, atelectasis, etc.), assessed by the researchers as unsuitable for inclusion 10. Acute cardiovascular and cerebrovascular accidents such as acute cerebral infarction, acute coronary syndrome, etc. within 3 months; 11. Subjects with severe cardiac dysfunction; history of severe arrhythmias in the past 2 years, including rapid atrial arrhythmias, any rapid ventricular arrhythmias; history of II degree type II or III degree atrioventricular block; and sinus bradycardia with a heart rate of less than 45 beats per minute, etc.; 12. Subjects have participated in or are participating in other clinical trials within three months; 13. Pregnant, lactating women, or women who plan to become pregnant during the study; 14. Subjects determined by the researchers to have other conditions that are unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
6-month complete ablation rate | 6 months

SECONDARY OUTCOMES:
Technical success rate | immediately after the PEF ablation treatment
6-month pulmonary progression-free survival rate | 6 months after the first PEF ablation treatment
12-month complete ablation rate | 12 months after the first PEF ablation treatment
12-month pulmonary progression-free survival rate | 12 months after the first PEF ablation treatment
  The proportion of subjects with no pulmonary progression (the first ablation lesion maintained no progression, no hilar lymph node metastasis, no new lesions) accounted for the proportion of evaluable subjects who received ablation
12-month overall survival rate | 12 months after the first PEF ablation treatment

OTHER OUTCOMES:
Safety of Intervention | 12 months
  All adverse events were recorded and evaluated according to CTCAE v5.0 (if applicable), and the relevance to the device itself and the treatment was evaluated. The incidence of device-related and surgical treatment-related adverse events and serious adverse events was calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine,, Shanghai, China